CLINICAL TRIAL: NCT07204639
Title: Safety and Efficacy of RAP-103 in Dose of 400mg/Day/One Dose a Day, 200mg/Day Twice Dose a Day, or Placebo Administrated for 8 Weeks, to Improve Severity and Quality of Life on Moderate to Severe Psoriasis in Subjects 18y to 70y: Randomized, Double Blind, Phase 2, Proof of Concept, Placebo Controlled Clinical Trial
Brief Title: Safety and Efficacy of RAP-103 to Improve Severity and Quality of Life on Moderate to Severe Psoriasis in Subjects
Acronym: RAP103-Pso
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Clarent Biopharma, Inc. (Industry)
Collaborators: Elemental Traslational Research SAPI (Unknown); Innovacion y Desarrollo de Estrategias en Salud (Other); Elemental CRO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAP103-202507-PoC
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis
Keywords: RAP103, Randomized trail phase 2, RAP103
MeSH Terms: conditions — Psoriasis | interventions — RAP-103; BID protein, human

STUDY DESIGN:
Intervention Model Description: Subjects will be included in 4 different parallel groups:
  * Group 1 to receive 400mg/day/oral/one dose a day of RAP-103 for 8weeks
  * Group 2 to receive 200mg/day/oral/twice dose a day of RAP-103 for 8weeks
  * Group 3 to receive Placebo for group for 400mg/day/oral/one dose a day 8weeks
  * Group 3 to receive Placebo for group for 200mg/day/oral/twice dose a day for 8weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RAP103 Active 400mg single dose (Experimental)
  Interventions: Drug: RAP103 400mg single dose
- RAP103 Active 200mg BID (Experimental)
  Interventions: Drug: RAP103 200mg BID
- Placebo for RAP 400mg (Placebo Comparator)
  Interventions: Drug: Placebo for RAP400
- Placebo for 200mg (Placebo Comparator)
  Interventions: Drug: Placebo for RAP200mg

INTERVENTIONS:
Drug: RAP103 400mg single dose — RAP103 400mg single dose, orally 8 weeks
  Arms: RAP103 Active 400mg single dose
Drug: RAP103 200mg BID — RAP103 200mg BID, orally 8 weeks
  Arms: RAP103 Active 200mg BID
Drug: Placebo for RAP400 — Placebo for RAP400mg single dose for 8 weeks
  Arms: Placebo for RAP 400mg
Drug: Placebo for RAP200mg — Placebo for RAP400mg single dose for 8 weeks
  Arms: Placebo for 200mg

SUMMARY:
Randomized, controlled trial, Proof of Concept, Phase 2 aimed to evaluate the effect of RAP-103 in dose of 400mg/day/one dose a day, 200mg/day twice dose a day, or placebo administrated for 8 weeks to improve Psoriasis Area and Severity Index (PASI)75 or static Physician's Global Assessment (sPGA) score of 0 or 1; PASI50, PASI90, PASI100, Scalp-specific Physician's Global Assessment (Ss-PGA) 0/1 with at least a 2-point improvement among patients with a baseline ss-PGA ≥3, sPGA 0, PSSD symptom score of 0 among patients with baseline score ≥1, Dermatology Life Quality Index (DLQI) 0/1 at Week 4 and 8 among patients with baseline DLQI ≥2, adjusted by transcriptomics profile (post-hoc analysis), Percentage of subjects which achieve The Minimum Clinically Important Difference (MCID) on DLQI (a ≥4-point reduction from baseline) at Week 4 and 8, Frequency of solicited and unsolicited adverse events (SAEs and USAEs) (Medra), and Changes on inflammatory and anti-inflammatory cytokine levels during treatment (IL-17, IL-23, IL-6, TNF-alpha, IL1-b, IL-10).

DETAILED DESCRIPTION:
Safety and Efficacy of RAP-103 in dose of 400mg/day/one dose a day, 200mg/day twice dose a day, or placebo administrated for 8 weeks, to improve severity and quality of life on moderate to severe psoriasis in subjects 18y to 70y: Randomized, double blind, phase 2, Proof of Concept, placebo controlled clinical trial. Primary Aim: To assess the effect over 8 weeks of oral RAP-103 (Dose 400mg/day/one dose a day, 200mg/day twice dose a day), or placebo on Psoriasis Area and Severity Index (PASI)75 or static Physician's Global Assessment (sPGA) score of 0 or 1; Secondary Aims: To assess the effect over 8 weeks of oral RAP-103 (Dose 400mg/day/one dose a day, 200mg/day twice dose a day), or placebo on secondary clinical improvement on PASI50, PASI90, PASI100, Scalp-specific Physician's Global Assessment (Ss-PGA) 0/1 with at least a 2-point improvement among patients with a baseline ss-PGA ≥3, sPGA 0, PSSD symptom score of 0 among patients with baseline score ≥1, Dermatology Life Quality Index (DLQI) 0/1 at Week 4 and 8 among patients with baseline DLQI ≥2, adjusted by transcriptomics profile (post-hoc analysis), Percentage of subjects which achieve The Minimum Clinically Important Difference (MCID) on DLQI (a ≥4-point reduction from baseline) at Week 4 and 8, Frequency of solicited and unsolicited adverse events (SAEs and USAEs) (Medra), and Changes on inflammatory and anti-inflammatory cytokine levels during treatment (IL-17, IL-23, IL-6, TNF-alpha, IL1-b, IL-10). Adults 18 years to 70y of age with moderate to severe plaque psoriasis who fulfill the inclusion criteria will be included in the study. Patients with a history of prior therapy, including biologic therapy, could be included after specified washout periods before randomization. Subjects will be included in 3 different groups: A) Group 1 to receive 400mg/day/oral/one dose a day of RAP-103 for 8weeks, B) Group 2 to receive 200mg/day/oral/twice dose a day of RAP-103 for 8weeks and C) Group 3 to receive Placebo for group for 400mg/day/oral/one dose a day 8weeks

o Group 3 to receive Placebo for group for 200mg/day/oral/twice dose a day for 8weeks. Throughout the trial, patients, investigators, and sponsors providing oversight remained blinded to treatment assignments. After completion of the 6-week period, eligible patients will be invited to enter to our full RCT phase 2, when they have at least 6 weeks without using RAP103 (washout period). The collection of nonserious AEs will start at initiation of study treatment until the final study visit. All SAEs will be collected from the date of the patient's written consent until 30 days after the final dose of the study drug or patient's participation in the study if the last scheduled visit occurred at a later time. The AEs of interest will include malignancies, infections (serious, opportunistic, fungal, tuberculosis, and herpes zoster), thromboembolic (arterial and venous) events, major adverse cardiovascular events (MACE; cardiovascular death, nonfatal myocardial infarction, and stroke), and skin events (acne and folliculitis). Solicited AEs will include select infection AEs, certain cardiovascular events, and suicidal ideation and behavior. All AEs will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA, version 28.0).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent

   a. Patients must be willing to participate in the study and sign the informed consent form
2. Type of patient and target disease characteristics

   1. Men and women, diagnosed with stable plaque psoriasis for 6 months or more. Stable psoriasis is defined as no morphology changes or significant flares of disease activity, in the opinion of the investigator
   2. Deemed by the investigator to be a candidate for systemic therapy
   3. ≥10% of body surface area (BSA) involvement at screening visit and Day 1
   4. Psoriasis Area and Severity Index (PASI) score ≥12, and static Physician's Global Assessment (sPGA) ≥3 at screening visit and Day 1
3. Age and reproductive status

   1. Men and women aged 18 years to 70 years at the time of screening visit
   2. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening visit, and a negative urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin within 24 hours prior to the start of study drug
   3. Women must not be pregnant, lactating, breastfeeding, or planning pregnancy during the study period
   4. Women of childbearing potential must agree to correctly use a highly effective method(s) of contraception for the duration of treatment plus 30 days (duration of ovulatory cycle) for a total of 33 days post-treatment completion (total of 33 days after last dose of study drug). WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements, but must still undergo pregnancy testing as described in this protocol
   5. Male patients who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment(s) plus 5 half-lives of the study treatment (3 days) for a total of 3 days post-treatment completion. Additionally, male patients must be willing to refrain from sperm donation during this time
   6. Investigators shall counsel WOCBP, and male patients who are sexually active with WOCBP, on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception, which have a failure rate of <1% when used consistently and correctly.

Exclusion Criteria:

1. Use of phototherapy 4 weeks or less prior randomization
2. Infectious/immune-related exclusions

   1. History or evidence of outpatient active infection and/or febrile illness within 7 days prior to Day 1
   2. History of serious bacterial, fungal, or viral infection requiring hospitalization and intravenous antimicrobial treatment within 60 days prior to Day 1
   3. Any untreated bacterial infection within 60 days prior to Day 1
   4. Any ongoing evidence of chronic bacterial infection (eg, chronic pyelonephritis, chronic osteomyelitis, chronic bronchiectasis)
   5. Any history of proven infection of a joint prosthesis in which the prosthesis was not removed or replaced, or received antibiotics for suspected infection of a joint prosthesis in which the prosthesis was not removed or replaced
   6. Received live vaccines within 60 days prior to Day 1, or plans to receive a live vaccine during the study, or within 60 days after completing study treatment
   7. Presence of herpes zoster lesions at screening or Day 1
   8. History of serious herpes zoster or serious herpes simplex infection, which includes, but is not limited to, any episode of disseminated herpes simplex, multidermatomal herpes zoster, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (recurrent is defined as 2 episodes within 2 years)
   9. Evidence of, or positive test for, hepatitis B virus at screening. Positive hepatitis B lab testing is defined as 1) positive hepatitis B surface antigen (HBsAg+) OR 2) presence of hepatitis B virus DNA OR 3) positive anti-hepatitis B core antibody without concurrent positive hepatitis B surface antibody (HBcAb+ and HBsAb-)
   10. Evidence of, or positive test for, hepatitis C virus (HCV) at screening. A positive test for HCV is defined as: positive for hepatitis C antibody (anti-HCV Ab) AND 2) positive via a confirmatory test for HCV (for example, HCV polymerase chain reaction)
   11. Positive for human immunodeficiency virus by antibody testing (HIV-1 and -2 Ab) at screening
   12. Any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the patient's immune status (eg, history of opportunistic infections [eg, Pneumocystis jirovecii pneumonia, histoplasmosis, or coccidioidomycosis], history of splenectomy, primary immunodeficiency)
3. Any of the following tuberculosis (TB) criteria:

   1. History of active TB prior to screening visit, regardless of completion of adequate treatment
   2. Signs or symptoms of active TB (eg, fever, cough, night sweats, and weight loss) during screening, as judged by the investigator
   3. Any imaging of the chest (eg, chest x-ray, chest computed tomography scan) obtained during the screening period, or any time within 6 months prior to screening with documentation, showing evidence of current active or history of active pulmonary TB
   4. Latent TB infection (LTBI) defined as positive interferon gamma release assay (IGRA), by QuantiFERON-TB Gold testing at screening, in the absence of clinical manifestations

   Note: Patient is eligible if (i) there are no current signs or symptoms of active TB AND (ii) patient has received adequate documented treatment for LTBI within 5 years of screening OR has initiated prophylactic treatment for LTBI per local guidelines and is rescreened after 1 month of treatment. To continue in the study, patient must agree to complete a locally recommended course of treatment for LTBI. Use of rifampin, however, is not recommended as it can reduce efficacy of apremilast used as a comparator in this trial

   Note: An IGRA test that is indeterminate must be retested for confirmation. If the second test is again indeterminate, the patient will be excluded from the study. If the retest is positive, the patient should be treated as having LTBI. If the retest is negative, the patient may be eligible provided no other exclusion criteria for TB are met.
4. Medical history and concurrent diseases

   1. Any major surgery within 8 weeks prior to Day 1, or any planned surgery for the first 52 weeks of the study
   2. Has donated blood >500 mL within 4 weeks prior to Day 1, or plans to donate blood during the course of the study
   3. Drug or alcohol abuse, as determined by the investigator, within 6 months prior to Day 1
   4. Medical marijuana or prescription marijuana taken for medicinal reasons
   5. Any major illness/condition or evidence of an unstable clinical condition (eg, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, psychiatric, neurologic, immunologic, or local active infection/infectious illness) that, in the investigator's judgment or after consultation with the medical monitor, will substantially increase the risk to the patient if he or she participates in the study
   6. Unstable cardiovascular disease, defined as a recent clinical cardiovascular event (eg, unstable angina, myocardial infarction, stroke, rapid atrial fibrillation) in the last 3 months prior to screening, or a cardiac hospitalization (eg, revascularization procedure, pacemaker implantation) within 3 months prior to screening
   7. Has uncontrolled arterial hypertension characterized by a systolic blood pressure (BP) >160 mm Hg or diastolic BP >100 mm Hg

      Note: Determined by 2 consecutive elevated readings. If an initial BP reading exceeds this limit, the BP may be repeated once after the patient has rested sitting for ≥10 minutes. If the repeat value is less than the criterion limits, the second value may be accepted.
   8. Class III or IV congestive heart failure by New York Heart Association Criteria
   9. Has cancer or history of cancer (solid organ or hematologic including myelodysplastic syndrome) or lymphoproliferative disease within the previous 5 years (other than resected cutaneous basal cell or squamous cell carcinoma, or carcinoma of cervix in situ that has been treated with no evidence of recurrence)
   10. Any uncontrolled psychiatric illness (such as untreated depression, or bipolar disorder) judged as clinically significant by the investigator during screening or at Day 1 OR any lifetime history of suicidal ideation, suicidal behavior, or suicidal attempts by medical history or by electronic Columbia-Suicide Severity Rating Scale (eC-SSRS) documentation, or by answering "yes" to Question 4 or 5 for suicidal ideation on the eC-SSRS at screening or at Day 1, or is clinically deemed to have a suicide risk by the investigator
   11. Prior exposure to investigational product on the last 6 months (ie, deucravacitinib or apremilast)
   12. If the patient has received biologics previously, the following exclusion criteria for washout will apply: Antibodies to IL-12, IL-17, or IL-23 (eg, ustekinumab, secukinumab, tildrakizumab, ixekizumab, or guselkumab) within 6 months of Day 1 prior randomization; Tumor necrosis factor inhibitor(s) (eg, etanercept, adalimumab, infliximab, certolizumab) within 2 months of Day 1; Agents that modulate integrin pathways to impact lymphocyte trafficking (eg, natalizumab), or agents that modulate B cells or T cells (eg, alemtuzumab, abatacept, or visilizumab) within 3 months of Day 1; or Rituximab within 6 months of Day 1
   13. Has received systemic nonbiologic psoriasis medications and/or any systemic immunosuppressant therapy (including, but not limited to, methotrexate, azathioprine, cyclosporine, Janus kinase inhibitors, 6-thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, tacrolimus, oral or injectable corticosteroids, retinoids, 1,25-dihydroxy vitamin D3 and analogues, psoralens, sulfasalazine, or fumaric acid derivatives) within 4 weeks prior to Day 1
   14. Has used leflunomide within 6 months prior to Day 1
   15. Has used opioid analgesics within 4 weeks prior to Day 1
   16. Has received lithium, antimalarials, or intramuscular gold within 4 weeks of the first administration of any study medication
   17. Has used any strong CYP450 inducers (eg, rifampin, phenobarbital, carbamazepine, phenytoin) within 4 weeks prior to Day 1
   18. Has used topical medications/treatments that could affect psoriasis evaluation (including, but not limited to, high potency corticosteroids (World Health Organization [WHO] Classes I-V), >3% salicylic acid, urea, alpha- or beta-hydroxyl acids, anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, methoxsalen, trimethylpsoralens, pimecrolimus, and tacrolimus) within 2 weeks prior to Day 1

       Note: Low-potency topical steroids (WHO Class VI and VII) are permitted on the palms, soles, face, and intertriginous areas but should not be used within 24 hours prior to any study visit. Bland emollients (defined as emollients without urea or alpha or beta hydroxy acids or other ingredients that are pharmaceutically active) are allowed on all body regions but should not be used within 24 hours prior to any study visit.
   19. Use of shampoos containing corticosteroids, coal tar, >3% salicylic acid, or vitamin D3 analogues within 2 weeks prior to Day 1
   20. Has received an experimental antibody or experimental biologic therapy within the previous 6 months OR received any other experimental therapy or new investigational agent within 30 days or 5 half-lives (whichever is longer) prior to Day 1 OR is currently enrolled in an investigational study
5. Laboratory evaluations

   1. Absolute white blood cell count <3000/mm3
   2. Absolute lymphocyte count <500/mm3
   3. Absolute neutrophil count <1000/mm3
   4. Platelet count <100,000/mm3
   5. Hemoglobin <9 g/dL
   6. Alanine aminotransferase and/or aspartate aminotransferase >3 × upper limit of normal (ULN)
   7. Total, unconjugated, and/or conjugated bilirubin >2 × ULN
   8. Thyroid-stimulating hormone outside the normal reference range AND free T4 (thyroxine) or T3 (triiodothyronine) outside the normal reference range
   9. Electrocardiogram abnormalities that are considered clinically significant and would pose an unacceptable risk to the patient if participating in the study
   10. Renal impairment based on an estimated glomerular filtration rate <45 mL/min

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-22 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index-75 | Day 0, Day 30 and Day 60
  Change on 75% at least for Psoriasis Area and Severity Index (PASI)75
static Physician's Global Assessment | Day 0, Day 30 and Day 60
  Change on static Physician's Global Assessment (sPGA) score of 0 or 1

SECONDARY OUTCOMES:
PASI50-100 | Day 0, Day 30 and Day 60
  Change on PASI50, PASI90, or PASI100 afetr treatment
Scalp-specific Physician's Global Assessment | Day 0, 30 and 60
  Change on Scalp-specific Physician's Global Assessment (Ss-PGA) 0/1 with at least a 2-point improvement among patients with a baseline ss-PGA ≥3
Psoriasis Symptoms and Signs Diary | Day 0, 30 and 60
  Changes on PSSD symptom score of 0 among patients with baseline score ≥1
Dermatology Life Quality Index | Day 0, 30 and 60
  Dermatology Life Quality Index (DLQI) 0/1 at Week 4 and 8 among patients with baseline DLQI ≥2
Frequency of adverse events | Day 30 and 60 after begin of treatment
  Frequency of solicited and unsolicited adverse events (SAEs and USAEs) (Medra)
Changes on inflammatory cytokines | Day 30 and 60 after treatment
  Changes on inflammatory and anti-inflammatory cytokine levels during treatment (IL-17, IL-23, IL-6, TNF-alpha, IL1-b, IL-10)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Narvaez Rosales, MD, Principal Investigator — Innovacion y Desarrollo de Estrategias en Salud
Locations (1):
- Innovacion y Desarrollo de Estrategias en Salud, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided